CLINICAL TRIAL: NCT04509414
Title: Intranasal Dexmedetomidine Versus Midazolam for Premedication in Deep-sedated Pediatric Dental Patients: a Double-blinded, Prospective, Randomized Controlled Trial
Brief Title: Intranasal Dexmedetomidine for Deep-sedated Pediatric Dental Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yang Xudong, Chief of Department of Anesthesiology, Peking University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PKUSSIRB-202056077
Record Dates: First submitted 2020-07-23; First posted 2020-08-12 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Deep Sedation; Dexmedetomidine
Keywords: deep sedation; pediatric; dexmedetomidine; dental treatment
MeSH Terms: interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dexmedetomidine (Experimental): 2ug/kg intranasal atomized dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- midazolam (Active Comparator): 0.2mg/kg intranasal atomized midazolam
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — For dexmedetomidine group after ramdomization, an intranasal dose of 2ug/kg dexmedetomidine will be administrated.
  Arms: dexmedetomidine
Drug: Midazolam — For midazolam group after ramdomization, an intranasal dose of 0.2mg/kg midazolam will be administrated.
  Arms: midazolam

SUMMARY:
It is important to choose an appropriate analgesia/sedation technique in pediatric dental treatment. Premedication combined with intravenous anesthesia is often used in deep sedation technique for pediatric dental treatment and it's a routine in most hospitals. Deep sedation has its unique advantages such as avoiding the airway damage with an enhanced recovery.

Dexmedetomidine is suitable for intranasal mucosal administration as a premedication drug. It has been proved with several beneficial characteristics in other clinical procedures.

This study intends to further explore the characteristics of nasal dexmedetomidine as premedication in pediatric oral treatment under deep sedation.

ELIGIBILITY:
Inclusion Criteria:

1. children in need of deep sedation for dental treatment aged 3-7 years.
2. anticipated operation time 1-2hours

Exclusion Criteria:

1. any known medical records with neural or mental disorder
2. any known medical records with severe systemic disorder
3. history of sedation drug administration in recent 1 months
4. any known allergic history of dexmedetomidine, midazolam or propofol
5. morbid obesity
6. history of OSAHS or acute respiratory infection in 2 weeks
7. other conditions which the attending considers to be unfit for the trial

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
venipuncture acceptance | Day 0
  acceptance while starting the IV line, at most 2 tries

SECONDARY OUTCOMES:
Observer's Assessment of Alertness/Sedation(MOAA/S) Score | Day 0
  sedation scoring with MOAA/S scale(from intranasal drug administration till discharge)
remedial mask induction acceptance | Day 0
  acceptance of the mask induction（for those failed to start the IV before induction）
propofol dosage | Day 0
  the total dosage of propofol used from induction till the end of the clinical treatment
patients' discomfort | up to 24 hours
  any adverse reaction or discomfort complaints of patients will be recorded, such as sneeze, blocked nose, bitter taste, dizziness, rhinalgia, etc.
hypoxemia | Day 0
  decreased oxygen saturation up to 90%, and the treatment will also be recorded(if any)
peri-operative blood pressure | Day 0
  peri-operative blood pressure states
peri-operative heart rate | Day 0
  peri-operative heart rate
times of intra-operative airway assistance | Day 0
  Any intra-operative airway assistance in need which aims to improve ventilation will be recorded, including jaw lifting, suction, mask ventilation and intubation. Specific type of assistance will also be recorded in detail.
post-operative pain | Day 0
  pain assessment with modified children's hospital of eastern Ontario pain score(m-CHEOPS) from the end of dental procedure till discharge
post-operative agitation | Day 0
  emergence agitation assessment with Pediatric Anesthesia Emergence Delirium scale(PAED) from the end of dental procedure till discharge
discharge time | Day 0
  time from the end of dental procedure till discharge

OTHER OUTCOMES:
peri-operative satisfaction | up to 24 hours
  satisfaction of surgeon and parents during the whole clinical treatment and follow-up, they will be asked to give a score from 1 to 10, 10 stands for completely satisfied and 1 stands for not satisfied at all
post-operative condition of the child | up to 24 hours
  complications and behavior changes assessed with Post-Hospitalization Behavior Questionnaire(PHBQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Hospital of Stomatology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided